CLINICAL TRIAL: NCT03855124
Title: The Effect of a Posture Shirt on Muscle Activity During Functional Tasks
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College of Northern Denmark (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor
Other Study IDs: FOU-UU-2018-12_Sub-project2
Record Dates: First submitted 2019-02-13; First posted 2019-02-26 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-02

CONDITIONS: Healthy
Keywords: Electromyography; Musculoskeletal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy participants: Participants will be ask to perform a repetitive upper limb task while posture and muscle activity is being monitored.This will be done while wearing a posture shirt or without a shirt
  Interventions: Device: Posture shirt

INTERVENTIONS:
Device: Posture shirt — Posture shirts are designed, and marketed to the general public and health service providers to improve posture and consequently alter muscle actitity, reduce musculoskeletal pain and discomfort.

SUMMARY:
This study sets out to investigate the effect of a posture shirt on muscle activity during a sitting and standing repetitive upper limb task

DETAILED DESCRIPTION:
Posture shirts are designed, and marketed to the general public and health service providers to improve posture and consequently alter muscle activity, reduce musculoskeletal pain and discomfort. This study sets out to investigate the effect of a posture shirt on muscle activity during a sitting and a standing repetitive upper limb task.

ELIGIBILITY:
Inclusion Criteria:

* Pain free healthy participants
* Able to speak, read and understand Danish

Exclusion Criteria:

* Pain from the back, neck or shoulder area during the past 6 months
* Experience of delayed onset muscle soreness (DOMS) on the day of testing
* Current or previous chronic or recurrent pain condition
* Regular use of analgesics
* Previous neurologic, musculoskeletal or mental illnesses that may influence the results
* Lack of ability to cooperate

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male participants
Study Population: healthy male participants
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-03-21 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Electromyography (EMG) | During the test session
  EMG acitivty of axioscapular and trunk muscles will be recorded during upper limb tasks

SECONDARY OUTCOMES:
Pain intensity: scale | During the test session
  Participants are to rate any perceived pain on a scale from 0-10 (0=no pain, 10= worst imaginable pain)

CONTACTS AND LOCATIONS:
Overall Officials: Steffan W Christensen, PhD, Principal Investigator — Department of Physiotherapy, University College of Northern Denmark
Locations (1):
- Department of Physiotherapy, University College of Northern Denmark, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided